CLINICAL TRIAL: NCT05717478
Title: Post-extraction Bone Regeneration of Partially Destroyed Sockets With Bovine Hydroxyapatite and rhBMP-2 Compared to Standard Guided Bone Regeneration Intervention (Bovine Hydroxyapatite and Collagen Membrane)
Brief Title: Regeneration of Alveolar Sockets With rhBMP-2-loaded Bovine Bone Mineral
Acronym: PROTEOGRAFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: NORICUM SL (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PIC-5-01; 894/21/EC-R (Other: Agencia Española del Medicamento y Productos Sanitarios (AEMPS)); CIV-ES-22-09-040949 (Other: European Data Base on Medical Devices (EUDAMED2))
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-01

CONDITIONS: Loss of Teeth Due to Extraction; Alveolar Bone Loss; Edentulous Alveolar Ridge
Keywords: Alveolar Bone Loss; Alveolar Ridge Augmentation; Bone Regeneration; Bone Morphogenetic Protein 2; Hydroxyapatite
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: Prospective and superiority therapeutic study with participants randomly distributed in two arms of equal size, one arm to receive Experimental treatment and the other Control treatment and blinded to participants and outcomes assessors.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Socket preservation after extraction with Proteo-Graft (Noricum S.L.) with a particle size of 0.25-1.00 mm, without using a barrier membrane.
  Interventions: Combination Product: rhBMP-2-BBM
- Control (Active Comparator): Conventional treatment (socket preservation therapy). Post-extraction socket preservation with Bio-Oss® (Geistlich Pharma AG, Switzerland) with a particle size of 0.25-1.00 mm, hereinafter BO, and protection with a barrier membrane, Bio-Gide® ( Geistlich Pharma AG, Switzerland).
  Interventions: Device: Bio-Oss+Bio-Gide

INTERVENTIONS:
Combination Product: rhBMP-2-BBM — Alveolar socket is filled with granules of bovine bone mineral (1.0-0.25 mm) loaded with human recombinant bone morphogenetic protein 2
  Arms: Experimental
Device: Bio-Oss+Bio-Gide — Alveolar socket is filled with granules of bovine bone mineral (Bio-Oss 1.0-0.25 mm) and covered with porcine collagen barrier membrane (Bio-Gide)
  Arms: Control

SUMMARY:
Aim of the present investigation will be to evaluate the efficacy and safety of a granulate of rhBMP-2- loaded bovine bone mineral (rhBMP-2-BBM) as alveolar bone regeneration procedure following tooth extraction.

Forty (40) patients (both sex; age 18 years and older) requiring extraction of one (1) hopeless tooth (incisor, canine or premolar with loss of bone height of 5 mm or more in buccal alveolar wall), followed by alveolar bone regeneration (ABR) and placement of an endosteal implant will be enrolled into the study.

After exodontia, participants will be randomized and divided into two groups: in Experimental Group the socket will be grafted with rhBMP-2-BBM granules (1.0-0.25 mm); in Control Group the sockets will be grafted with Bio-Oss granules (1.0-0.25 mm) and covered with porcine collagen barrier membrane (Bio-Gide).

The end of the study will be fixed at the implantation surgery, seventeen (17) weeks after exodontia an ABR. Cone beam computed tomography (CBCT) scans will be made, immediately after (0), and sixteen (16) weeks after exodontia an ABR and the gain in alveolar bone height will be estimated and used as the primary outcome for comparison of both groups.

As secondary efficacy outcomes the change in alveolar bone width estimated from the CBCT scans; initial (0) and at seventeenth (17th) week after tooth extraction; the change in dental arch dimensions estimated from tridimensional models obtained from intraoral scans at one week before (-1) and sixteen (16) weeks exodontia an ABR; and the amounts of new bone, remnant material and connective tissue histomorphometrically measured in a bone biopsy collected during the implantation surgery at seventeenth (17th) week, will be considered.

Healing of gingival tissues at first (1st) and second (2nd) week and incidence of adverse reactions at first (1st), second (2nd) and sixteenth (16th) week, are used as secondary safety outcomes.

DETAILED DESCRIPTION:
It is an interventional and therapeutic clinical trial, as well as unicentric, prospective, parallel, controlled, random, and doble-blind (participants and outcomes assessors).

It is aimed to assess the efficacy and safety of an experimental combined medical device consisting of rhBMP-2-loaded bovine bone mineral (rhBMP-2-BBM) granules (1.0-0.25 mm) for alveolar bone regeneration (ABR) after extraction of a hopeless tooth (incisor, canine or premolar, both in upper and lower arch maxilla), having not less than 5 mm of bone height loss in vestibular wall, and planned insertion of an endosteal dental implant and prosthetic rehabilitation.

Participants will be recruited among patients attending the Dental Clinic of the Faculty of Dentistry of the Universidad Complutense de Madrid, Spain. There will be enrolled forty (40) voluntary (both sex; age 18 years and older) requiring extraction of one (1) hopeless tooth (incisor, canine or premolar with loss of bone height of five (5) mm or more in vestibular alveolar wall), followed by alveolar bone regeneration (ABR) and placement of an endosteal implant. Participants will be randomly and equitably distributed in two groups; Experimental and Control, each counting 20 participants.

Experimental group will be treated with rhBMP-2-BBM granules (1.0-0.25 mm) and Control group with Bio-Oss granules (1.0-0.25 mmm) and porcine collagen barrier membrane (Bio-Gide).

The enrollment will be open a maximum period of 12 months. Treatment and follow-up will last 18 weeks between the enrollment of one participant and the end of the study.

The research hypothesis is "(rhBMP-2-BBM) is more effective than and as safe as Bio-Oss+Bio-Gide for ABR of post-exodontia sockets with severe loss of vestibular bone height."

Outcomes are:

* Primary Efficacy Outcome: Bone height gain 16 weeks after baseline, radiographically measured.
* Secondary Efficacy Outcomes:

  * Bone width change 16 weeks after baseline, radiographically measured.
  * Dental arch dimensional change 16 weeks after baseline, measured from digital models.
  * Need for second bone augmentation 17 weeks after baseline, clinically assessed.
  * Amounts of New Bone; Remnant Material and Connective Tissue 17 weeks after baseline, histomorphometrically measured.
* Secondary Safety Outcomes:

  * Early Healing Index 1 and 2 weeks after baseline, clinically assessed.
  * Adverse reactions 1, 2 and 16 weeks after baseline, clinically assessed. Enrollment: Potential participants will be asked and examined to check they fulfil the inclusion criteria and vestibular bone height of the affected tooth will be measured by probing. Those fulfilling inclusion criteria will receive detailed explanation on the characteristics of the trial, their rights as participant, and asked for their consent to participate. Those accepting will receive a copy of the informed consent form, and will be scheduled for a First Visit.

First Visit (1 week before baseline): Participants will be asked to confirm full comprehension of their rights and duties and their will to participate, and required to provide the signed informed consent form. A digital scan of affected area including hopeless tooth and it neighbors will be obtained. The resulting STL file will be used to obtain the base dimensional measure of the alveolar ridge. The base STL file will be also used to design a customized splint which will be manufactured in thermoplastic polymer by 3D-printing and used in all CBCT scans to standardize radiographic measurements of height and width of the alveolar bone. The Second Visit will be scheduled in the term of 1 week (± 1 day) and participant will be indicated to brush teeth thrice a day and to rinse mouth with 0.12 % chlorhexidine twice a day till the appointment day, and amoxicillin 750 mg/8 h (or clindamycin 300 mg/6 h) for 24 h before the appointment day.

Second Visit (baseline): Atraumatic exodontia will be carried out under local anesthesia using a syndesmotome, manual or coupled to a piezosurgery unit, avoiding to damage the alveolar bone walls. The vestibular bone height will be probed to confirm the loss is greater than 5 mm. If not, the patient will be excluded and will continue to be treated by conventional procedures. Socket will be thoroughly curetted and CBCT scan with the customized splint will be obtained before the ABR treatment. Treatment with rhBMP-2-BBM or Bio-Oss+Bio-Gide will be randomly assigned and ABR procedure will be performed.

The socket is to be filled to the height of the interdental bone tables with the granules and gingiva is sutured with cross mattress stitches. For control group the granules of Bio-Oss will be covered with the Bio-Gide membrane before suturing.

The Third Visit will be scheduled in the term of 1 week (± 2 days) and amoxicillin 750 mg/8 h (or clindamycin 300 mg/6h horas) during the next 8 days is to be indicated; acetaminophen 1 g/8 h (in case of pain) and ibuprofen 400 mg/8 h (in case of swelling) till remission of symptoms. Oral care for the next two (2) weeks will consist in normal teeth brushing excluding the affected area, mouth rinsing with 0.12 % chlorhexidine twice a day, and avoiding use any removable prosthesis affecting regenerated area. A phone number will be provided to report any persistent (4-5 days) adverse effect or emergency.

Third Visit (1 week after baseline): Healing and adverse reactions outcomes will be assessed. The Early Healing Index (PMID: 12795787) will be used for healing assessment. Adverse reactions are to be assessed on the basis of clinical exam and participant questioning. Reactions to consider are facial erythema, local edema, local erythema; fever; local pain; granules exfoliation, and suppuration; and will be qualified as none, mild, moderate, or severe. A unique blind outcome assessor previously trained will assess both outcomes. Stitches will be removed and the Fourth Visit scheduled in a term of 2 weeks (±2 days) from baseline.

Fourth Visit (2 weeks after baseline): Assessment of healing and adverse reactions outcomes will be performed as above and the Fifth Visit will be scheduled in a term of 16 weeks (±1 week) after baseline.

Fifth Visit (16 weeks after baseline):

Clinical exam and assessment of adverse reactions outcome will be performed. Digital and CBCT (using the customized splint) scans will be obtained and used to assess the outcomes of bone height gain and bone width change according to (PMID: 30883942) and dental arch dimensional change as stated by (PMID: 30508313) by trained and calibrated blind assessor. The Sixth Visit will be scheduled in the term of 17 weeks (± 1 week) and participant will be indicated as in the first visit.

Sixth Visit (17 weeks after baseline, End of Study): A buccal full thickness flap will be elevated and dimensions and quality of the alveolar bone ridge will be inspected to assess the need for second bone augmentation outcome. If second bone augmentation is needed, participant goes out the trial, receive the bone augmentation and continues conventional treatment.

If no need for second bone augmentation, a biopsy specimen of the alveolar regenerated bone will be harvested exactly in the area where dental implant will be placed. At this point, participant exit the study and goes on to conventional endosteal implantation and subsequent prosthetic rehabilitation.

The biopsy specimen is fixed in 10 % buffered formalin and kept at 4 ºC until processing for histology and histomorphometry studies (PMID: 6809919). The amounts of New Bone; Remnant Material and Connective Tissue 17 weeks after baseline will be assessed by a trained and calibrated blind assessor as indicated in (PMID: 28634845).

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients with one tooth to be extracted, from incisor to premolar, and with buccal bone wall loss of 5 mm or more
* Plaque index lower than 30%
* Eighteen (18) years old and elder.
* Willing to participate and written informed consent

Exclusion Criteria:

* Heavy smokers (more than 20 cigarettes per day)
* Plaque index greater than 30 %
* Pathologies hindering interventions or influencing healing or host response
* Inability to comply scheduled follow-up
* Comprehension disability that compromises informed consent and compliance with medical instructions
* Receptor of any other experimental treatments, actual or in past 30 days
* Current pregnant patients or planning to get pregnant in short term
* Breastfeeding mothers

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Bone height gain after tooth extraction and socket regeneration | 16 weeks
  Difference between alveolar bone heights measured immediately after tooth extraction and 16 weeks after. Bone heights are measured from the CBCT scans obtained in the second and fifth visits using as reference a customized splint as elsewhere (PMID: 30883942)

SECONDARY OUTCOMES:
Bone width changes after tooth extraction and socket regeneration | 16 weeks
  Difference between alveolar bone widths measured immediately after tooth extraction and 16 weeks after. Bone widths are measured at 25%, 50% and 75% of bone height from the CBCT scans obtained in the second and fifth visits using as reference a customized splint as elsewhere (PMID: 30883942)
Dental arch dimensional changes after tooth extraction and socket regeneration | 16 weeks
  Differences between volumes and widths of the dental arch region affected measured 1 week before and 16 weeks after tooth extraction. Arch widths are measured at distances of 1, 2, 3, 4 and 5 mm from gingival margin. Digital models of the affected area obtained from the intraoral scans obtained in the first and fifth visits are used for measures as elsewhere (PMID: 30508313)
Need for second bone augmentation after tooth extraction and socket regeneration | 17 weeks
  The outcome will be intraoperatively assessed at the surgery of Sixth Visit after rising buccal full thickness flap and exposing the regenerated area. The outcome assessor will exam the regenerated socket and will decide if the quality and volume of bone is enough to continue to the insertion of a endosteal implant (NO); or further bone augmentation is needed (YES)
Amounts of New Bone; Remnant Material and Connective Tissue after tooth extraction and socket regeneration | 17 weeks
  At the surgery of the Sixth Visit a biopsy of the alveolar regenerated bone will be harvested exactly in the place where endosteal implant is to be inserted, with the aid of a trephine bur. The bur with the specimen is fixed in formalin, dehydrated and resin embedded. Longitudinal sections will be cut and polished and dyed with Levai-Laczkó stain (PMID: 68009919) and the percentages of New Bone; Remnant Material and Connective Tissue will be histomorphometrically measured as elsewhere (PMID: 28634845)
Early Healing Index after tooth extraction and socket regeneration | 1 and 2 weeks
  At the clinical exam in Third and Fourth Visits the outcome assessor will qualify the Early Healing Index using a scale of 1 to 5 as elsewhere (PMID: 12795787)
Adverse reactions after tooth extraction and socket regeneration | 1, 2 and 16 weeks
  Adverse reactions will be assessed on the basis of clinical exam and participant questioning practiced by the outcome assessor at Third, Fourth and Fifth Visits. Reactions to consider are: facial erythema, local edema, local erythema, fever, local pain, granules exfoliation, and suppuration; and they will be qualified as none, mild, moderate, or severe. Any other reaction observed will be registered and qualified with the same scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sanz, MD,PHD, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Faculty of Dentistry, Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wachtel H, Schenk G, Bohm S, Weng D, Zuhr O, Hurzeler MB. Microsurgical access flap and enamel matrix derivative for the treatment of periodontal intrabony defects: a controlled clinical study. J Clin Periodontol. 2003 Jun;30(6):496-504. doi: 10.1034/j.1600-051x.2003.00013.x. PMID 12795787
- [Background] Jo DW, Cho YD, Seol YJ, Lee YM, Lee HJ, Kim YK. A randomized controlled clinical trial evaluating efficacy and adverse events of different types of recombinant human bone morphogenetic protein-2 delivery systems for alveolar ridge preservation. Clin Oral Implants Res. 2019 May;30(5):396-409. doi: 10.1111/clr.13423. Epub 2019 Apr 11. PMID 30883942
- [Background] Sanz-Martin I, Encalada C, Sanz-Sanchez I, Aracil J, Sanz M. Soft tissue augmentation at immediate implants using a novel xenogeneic collagen matrix in conjunction with immediate provisional restorations: A prospective case series. Clin Implant Dent Relat Res. 2019 Feb;21(1):145-153. doi: 10.1111/cid.12696. Epub 2018 Dec 3. PMID 30508313
- [Background] Donath K, Breuner G. A method for the study of undecalcified bones and teeth with attached soft tissues. The Sage-Schliff (sawing and grinding) technique. J Oral Pathol. 1982 Aug;11(4):318-26. doi: 10.1111/j.1600-0714.1982.tb00172.x. PMID 6809919
- [Background] Ortiz-Vigon A, Martinez-Villa S, Suarez I, Vignoletti F, Sanz M. Histomorphometric and immunohistochemical evaluation of collagen containing xenogeneic bone blocks used for lateral bone augmentation in staged implant placement. Int J Implant Dent. 2017 Dec;3(1):24. doi: 10.1186/s40729-017-0087-1. Epub 2017 Jun 21. PMID 28634845